CLINICAL TRIAL: NCT04788576
Title: Distribution and Clinical Implication of Coronary Flow Reserve and Index of Microcirculatory Resistance in Patients With Heart Failure With Preserved Ejection Fraction Without Significant Coronary Artery Disease
Brief Title: Distribution and Clinical Implication of CMD in Patients With HFpEF Without Significant CAD
Acronym: HFpEF-CMD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Ki Hong Choi, Clinical Assistant Professor, Samsung Medical Center
Other Study IDs: HFpEF_CMD
Record Dates: First submitted 2021-03-05; First posted 2021-03-09 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Heart Failure With Preserved Ejection Fraction; Coronary Microvascular Dysfunction
Keywords: Heart failure with preserved ejection fraction; Coronary physiology; Coronary microvascular dysfunction; HFA-PEFF score

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with heart failure with preserved ejection fraction (HFpEF): Subject with preserved ejection fraction (ejection fraction > 50%) and with dyspnea on exertion (NYHA Grade 2 or more) and diagnosed as HFpEF using HFA-PEFF scoring system (HFA-PEFF ≥5 or 2-4 with abnormal stress test or invasive hemodynamic test)
  Interventions: Diagnostic Test: Invasive physiologic evaluation (fractional flow reserve, coronary flow reserve, index of microcirculatory resistance)

INTERVENTIONS:
Diagnostic Test: Invasive physiologic evaluation (fractional flow reserve, coronary flow reserve, index of microcirculatory resistance) — In case of heart failure with preserved ejection fraction confirmed by HFA-PEFF scoring system without functionally significant coronary artery disease, coronary angiography with invasive physiologic evaluation including fractional flow reserve, coronary flow reserve, and index of microcirculatory resistance will be performed to evaluate the distribution and clinical implication of coronary microvascular dysfunction.

SUMMARY:
To evaluate the incidence of coronary microvascular dysfunction (CMD) and its' prognostic implication in patients who have diagnosed as heart failure with preserved ejection fraction (HFpEF) confirmed by HFA-PEFF scoring system without functionally significant coronary artery disease.

DETAILED DESCRIPTION:
Heart failure with preserved ejection fraction (HFpEF) is a clinical syndrome in patients with current or prior symptoms of HF with a left ventricular ejection fraction (LVEF) ≥ 50 percent and evidence of cardiac dysfunction as a cause of symptoms (abnormal LV filling and elevated filling pressures). Previous studies have reported that HFpEF is related to various clinical risk factors such as hypertension, obesity, diabetes mellitus, chronic kidney disease, atrial fibrillation, myocardial ischemia with or without significant epicardial coronary artery stenosis, or myocardial infiltrative disease. Although its pathophysiology remains incompletely understood, findings from clinical and pre-clinical studies have suggested systemic endothelial dysfunction, oxidative stress, and coronary microvascular dysfunction (CMD) could be important pathophysiologic mechanisms for HFpEF.

In this regard, recent studies evaluated non-invasively measured coronary flow reserve (CFR) from positron emission tomography (PET), cardiac magnetic resonance imaging (MRI), or Doppler echocardiography, and presented the association of depressed global CFR with cardiac diastolic dysfunction and higher risk of clinical events. The presence of CMD can be also evaluated by invasive physiologic assessment using both CFR and index of microcirculatory resistance (IMR). Nevertheless, there has been limited study which evaluated the association between HFpEF and CMD using invasive physiologic indices and their prognostic implications, especially in patients without significant coronary artery stenosis. Therefore, we sought to evaluate the incidence of CMD and its' prognostic implication in patients who have diagnosed as heart failure with preserved ejection fraction (HFpEF) confirmed by HFA-PEFF scoring system without functionally significant coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be at least 19 years of age.
* Subject with preserved ejection fraction (ejection fraction > 50%)
* Subject presented with dyspnea on exertion (NYHA Grade 2 or more) and diagnosed as HFpEF using HFA-PEFF scoring system (HFA-PEFF ≥5 or 2-4 with abnormal stress test or invasive hemodynamic test)
* Subject who clinically need coronary angiography
* Subject who is able to voluntarily sign informed consent form

Exclusion Criteria:

* Subject with reduced ejection fraction (<50%)
* Subject with significant coronary artery stenosis on coronary angiography (diameter stenosis ≥90% or 50-90% with fractional flow reserve [FFR] ≤0.80)
* Subject who has other obvious causes of dyspnea (ex, lung disease)
* Subject who have non-cardiac co-morbid conditions with life expectancy <1 year

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have diagnosed as heart failure with preserved ejection fraction (HFpEF) confirmed by HFA-PEFF scoring system without functionally significant coronary artery disease
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-01-25 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of CMD in patients with HFpEF | Immediate after the index procedure
  Proportion of CMD confirmed by invasive physiologic evaluation

SECONDARY OUTCOMES:
Correlation between CMD and left ventricular end diastolic pressure | Immediate after the index procedure
  Correlation between CMD confirmed by invasive physiologic evaluation and left ventricular end diastolic pressure
Correlation between CMD and E/e' | Immediate after the index procedure
  Correlation between CMD confirmed by invasive physiologic evaluation and E/e'
Correlation between CMD and HFA-PEFF score | Immediate after the index procedure
  Correlation between CMD confirmed by invasive physiologic evaluation and HFA-PEFF score
Correlation between CMD and NT-proBNP | Immediate after the index procedure
  Correlation between CMD confirmed by invasive physiologic evaluation and NT-proBNP
Correlation between CMD and pulmonary artery wedge pressure | Immediate after the index procedure
  Correlation between CMD confirmed by invasive physiologic evaluation and pulmonary artery wedge pressure
Correlation between CMD and mean pulmonary artery pressure | Immediate after the index procedure
  Correlation between CMD confirmed by invasive physiologic evaluation and mean pulmonary artery pressure
All-cause death | At 2 years after the index procedure
  All-cause death during follow-up
Cardiac death | At 2 years after the index procedure
  Cardiac death during follow-up
Myocardial infarction | At 2 years after the index procedure
  Myocardial infarction during follow-up
Any revascularization | At 2 years after the index procedure
  Any revascularization during follow-up
Readmission due to heart failure | At 2 years after the index procedure
  Readmission due to heart failure during follow-up
Readmission | At 2 years after the index procedure
  Readmission during follow-up
Proportion of heart failure with reduced ejection fraction | At 2 years after the index procedure
  Proportion of progression of heart failure with reduced ejection fraction
Correlation between CMD and Excercise induced E/e' | Immediate after the index procedure
  Correlation between CMD confirmed by invasive physiologic evaluation and exercise induced E/e'
Correlation between CMD and Exercise induced pulmonary artery wedge pressure | Immediate after the index procedure
  Correlation between CMD confirmed by invasive physiologic evaluation exercise induced and pulmonary artery wedge pressure
Correlation between CMD and exercise time | Immediate after the index procedure
  Correlation between CMD confirmed by invasive physiologic evaluation exercise time
Correlation between CMD and mean exercise induced pulmonary artery pressure | Immediate after the index procedure
  Correlation between CMD confirmed by invasive physiologic evaluation and exercise induced mean pulmonary artery pressure
Correlation between CMD and Gas analysis data (Peak exercise oxygen consumption, Respiratory quotient) | Immediate after the index procedure
  Correlation between CMD confirmed by invasive physiologic evaluation and exercise induced peak exercise oxygen consumption, Respiratory quotient

CONTACTS AND LOCATIONS:
Overall Officials: Ki Hong Choi, MD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea